CLINICAL TRIAL: NCT06866236
Title: Use of NAD Oxidase Modulation Agent QRX3 for Prevention and Treatment of Progressive Chronic Kidney Disease
Brief Title: Use of New Drug QRX-3 for Prevention and Treatment of Chronic Kidney Disease Progression
Acronym: NAD agent
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ebima Clifford Okundaye (Industry)
Responsible Party: Sponsor-Investigator, Ebima Clifford Okundaye, President, Neukidney Inc.
Organization: Neukidney Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Diseases; Acute Kidney Injury; Kidney Failure
Keywords: CKD, CKD treatment , renal function
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized placebo double control
Who Masked: Investigator
Masking Description: placebo arm with intervention pill arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Active Comparator): QRX-3 - two capsules orally twice daily
  Interventions: Drug: QRX-3
- placebo (Placebo Comparator): placebo pill - one capsule orally twice daily
  Interventions: Drug: QRX-3

INTERVENTIONS:
Drug: QRX-3 — capsule

SUMMARY:
Chronic kidney disease CKD is estimated to affect nearly over 800 million people globally today (with roughly 125,000 people ending up annually on dialysis in the United States alone. CKD is a contributor to illness and is associated with a diminished quality of life and reduced life expectancy . In this study the investigators are using a novel drug to target improved function of the kidneys.

DETAILED DESCRIPTION:
Chronic kidney disease has been linked to impaired activity of mitochondrial dysfunction along with oxidative intracellular mechanisms that result in the cascade of progressive damage within renal tubular cells. Several treatment options for mitochondrial dysfunction have been suggested to target the loss of nephrons via renal fibrosis and tubular senescence of the kidney cells by enhancing the mitochondrial activity of these cells via the NAD/NAD+ redox pathway as well as reduce the presence of fibrogenic intracellular inflammatory markers .

QRX-3 is a formulated novel drug designed to supply and optimize NAD+ mitochondrial availability and prevent this nephron loss .

In this study the investigators will evaluate the effect of intervention with this novel drug therapy on chronic kidney disease CKD population with slowly declining renal function.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  * Patient with Chronic kidney disease
  * Estimated Glomerular function by MDRD of less than 60mls/min
  * Patients with declining renal function ( as measured by eGFR by MDRD )
  * Rate of decline of eGFR over the last one year of less than 20%
  * Negative Serology markers for CKD etiology
  * Provider perceived adherence to study follow up

Exclusion Criteria:

Rapid rate of decline in kidney function of > 20 % over last one year

* Symptomatic renal failure
* Presence of any suspected Acute renal failure superimposed
* Presence of cast , hematuria, or abnormal urinalysis outside of simple UTI
* No known reversible cause of renal decline

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
change in Glomerular filtration rate | 1 year
  change percentage in kidney function level measured with cystatin creatinine glomerular filtration rate

SECONDARY OUTCOMES:
change in Proteinuria | 1 year
  change in random urine protein/creatinine ratio
change in rate of Glomerular filtration rate decline | 1 year
  comparism of slopes of decline in cystatin creatinine glomerular filtrate rate

CONTACTS AND LOCATIONS:
Locations (1):
- Neukidney Inc, Pasedena, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified information of each participants trial characteristics will be available for sharing